CLINICAL TRIAL: NCT02975622
Title: Immediate Complications According to Ultrasound-guided Central Venous Catheters Insertion Site: a Non-inferiority Randomized Clinical Trial Comparing Jugular and Subclavian Approaches
Brief Title: Immediate Complications According to Ultrasound-guided Central Venous Catheters Insertion Site: a Non-inferiority Randomized Clinical Trial
Acronym: USCATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Jose Augusto Santos Pellegrini, MD, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCPA001
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Catheterization, Central Venous; Ultrasonography
MeSH Terms: interventions — Catheterization, Central Venous

ARMS (2):
- Subclavian (Active Comparator): Subclavian vein will be individualized and approached by longitudinal incidence, according to previous studies. Skin puncture will be made next to the transducer, lateral to the first rib, maintaining constant visualization of the needle tip.
  Interventions: Procedure: Central venous catheterization
- Jugular (Active Comparator): Jugular vein will be identified by transverse or longitudinal approach, and skin puncture will be made by transverse or longitudinal incidence, according to operator's preferences. Using transverse approach, the needle will be maintained in a 45 degree angle with the skin, and the insertion site will be exactly the same as the measured distance between asking and jugular vein wall.
  Interventions: Procedure: Central venous catheterization

INTERVENTIONS:
Procedure: Central venous catheterization — Ultrasound guided central venous catheterization

SUMMARY:
Ultrasound (US)-guided central venous catheterization is now considered standard of care according to recent clinical evidence, at least considering jugular vein approach. Recent trials suggested that even US-guided subclavian approach could be more effective that landmark technique. However, studies comparing both sites employing US are still lacking.

We, therefore, designed a non-inferiority randomized controlled trial to compare these sites, both using US guidance, according to immediate complications following central venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients; central venous access indicated.

Exclusion Criteria:

* cardiac arrest; at least one side of each vein available for insertion; pacemaker insertion; pulmonary artery catheter insertion; non-corrected coagulopathy; thrombolytics in the past 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Immediate complications | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil